CLINICAL TRIAL: NCT07080398
Title: The Utility of Transcutaneous Bilirubin Measurement in Term and Late-Preterm Infants With Hyperbilirubinemia: A Prospective Observational Study During and After Phototherapy
Brief Title: Accuracy of TcB Measurements During and After Phototherapy
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Seda Yilmaz Semerci, Assoc. Prof., Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: 2021/249
Record Dates: First submitted 2025-07-15; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Neonatal Hyperbilirubinemia
Keywords: newborn; hyperbilirubinemia; phototherapy; bilirubin; transcutaneous bilirubin; serum bilirubin
MeSH Terms: conditions — Hyperbilirubinemia, Neonatal; Hyperbilirubinemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Biospecimen Retention: Samples Without DNA — Serum bilirubin level
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- term newborns: term newborns with hyperbilirubinemia requiring phototherapy
  Interventions: Diagnostic Test: serum bilirubin level measurement
- late-preterm newborns: late-preterm newborns with hyperbilirubinemia requiring phototherapy
  Interventions: Diagnostic Test: serum bilirubin level measurement

INTERVENTIONS:
Diagnostic Test: serum bilirubin level measurement — Total serum bilirubin levels and concurrent transcutaneous bilirubin measurements will be done and the results will be evaluated comperatively.

SUMMARY:
This study aimed to assess the accuracy of transcutaneous bilirubin measurements in term and late-preterm infants undergoing phototherapy. Transcutaneous bilirubin levels were measured from different anatomical sites during and after treatment, and compared to total serum bilirubin levels. The agreement between the two methods was evaluated using Bland-Altman plots.

DETAILED DESCRIPTION:
This study focused on evaluating the accuracy of transcutaneous bilirubin measurements in term and late-preterm infants who were receiving phototherapy treatment. Transcutaneous bilirubin levels were measured at two different locations - the glabella (forehead) and lower abdomen - while the infants were undergoing phototherapy. These measurements were then compared to total serum bilirubin levels, which is the gold standard for assessing bilirubin levels in the blood.

The researchers used Bland-Altman plots to analyze the agreement between the transcutaneous bilirubin measurements and total serum bilirubin levels.

By comparing the transcutaneous bilirubin measurements to total serum bilirubin levels using Bland-Altman plots, the researchers were able to determine the accuracy of the transcutaneous measurements in this specific population of infants undergoing phototherapy. This information is important for healthcare providers to ensure that they are using the most accurate and reliable method for monitoring bilirubin levels in infants receiving treatment for jaundice.

ELIGIBILITY:
Inclusion Criteria:

* Newborn infants less than 7 days of life
* Hyperbilirubinemia requiring phototherapy
* Indirect hyperbilirubinemia
* Newborn infants who are born between 35-42 weeks of gestation

Exclusion Criteria:

* Direct hyperbilirubinemia
* Disease states other than hyperbilirubinemia
* Congenital abnormalities
* Chromosomal abnormalities
* Poor peripheral perfusion
* Edema

Ages: 1 Hour to 2 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Term and late-preterm newborn infants with hyperbilirubinemia requiring photothrepy will be included.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Correlation coefficient of transcutaneous bilirubin (TcB) and total serum bilirubin (TSB) | from enrollment to 24th hour after the end of the phototherapy treatment
  The accuracy of TcB as a substitute of TSB will be evaluated through correlation and Bland-Altman analysis

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences Istanbul KSS Training and Research Hospital, Istanbul, Kucukcekmece, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
can be shared after the study is published.